CLINICAL TRIAL: NCT04417725
Title: Burden of Disease of Chronic Kidney Disease (CKD), Type 2 Diabetes Mellitus (T2DM), and Comorbid T2DM/CKD in Alberta, Canada: A Non-interventional Study Using Administrative Health Data
Brief Title: Burden of Chronic Kidney Disease (CKD), Type 2 Diabetes Mellitus (T2DM), and Comorbid T2DM/CKD in Alberta, Canada
Status: Completed | Type: Observational
Sponsor: Medlior Health Outcomes Research Ltd (Other)
Responsible Party: Principal Investigator, Tara Cowling, Director and Managing Principal, Medlior Health Outcomes Research Ltd
Other Study IDs: 1245.217
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Diseases; Type 2 Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic kidney disease: Adult patients (≥18 years of age) with CKD were identified in Alberta during the case ascertainment period (April 1, 2010, to March 31, 2019), based on a validated algorithm incorporating ICD-9-CM/ICD-10-CA coding, estimated glomerular filtration rate, and albuminuria laboratory tests. This is a non-interventional, observational study, and thus, no intervention was administered.
  Interventions: Other: Not applicable - this is a non-interventional, observational study.
- Type 2 diabetes mellitus: Adult patients with T2DM were identified in Alberta during the case ascertainment period (April 1, 2010 to March 31, 2018), based on a validated algorithm incorporating ICD-9-CM and ICD-10-CA codes. This is a non-interventional, observational study, and thus, no intervention was administered.
  Interventions: Other: Not applicable - this is a non-interventional, observational study.
- Comorbid type 2 diabetes mellitus and chronic kidney disease: The derived T2DM cohort was used to identify patients with comorbid T2DM/CKD (stages 1-3) during the same case ascertainment period (April 1, 2010 to May 31, 2018). The study cohort included T2DM patients with comorbid CKD (stages 1-3) identified in Alberta within the two years prior or after their T2DM index date, using the T2DM index date as the index date for this cohort. This is a non-interventional, observational study, and thus, no intervention was administered.
  Interventions: Other: Not applicable - this is a non-interventional, observational study.

INTERVENTIONS:
Other: Not applicable - this is a non-interventional, observational study. — Not applicable - this is a non-interventional, observational study.

SUMMARY:
The purpose of the research study is to describe the burden of disease among three different cohorts of patients: (1) patients diagnosed with CKD, (2) those with T2DM; and (3) those with T2DM and comorbid CKD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) has been ranked as the 10th leading cause of death in Canada as of 2013, while type 2 diabetes mellitus (T2DM) is one of the fastest growing diseases in Canada. There is a growing body of evidence that has examined these populations in real-world settings in Canada. The study described below will add to the growing body of literature that has examined CKD patients in Alberta and will contribute to an understanding of the epidemiology of CKD by stage, as well as healthcare resource utilization (HCRU) and costs. Furthermore, this study will contribute to a more nuanced understanding of the epidemiology, treatment patterns, HCRU and costs, and adverse events for T2DM patients with and without comorbid CKD in Alberta.

ELIGIBILITY:
Inclusion Criteria (either of the following):

* Chronic kidney disease identified using laboratory test and health administrative data
* Type 2 diabetes mellitus identified using health administrative data

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD will be defined using a published algorithm based on ICD-9-CM/ICD-10-CA diagnostic codes and eGFR/albuminuria laboratory test values.
  Patients with T2DM will be defined using a published algorithm based on ICD-9-CM/ICD-10-CA diagnostic codes.
  Patients with comorbid T2DM/CKD will be identified among patients identified with prevalent T2DM. CKD comorbidity will be defined as identified CKD within the two years prior or any time after the T2DM index date.
Sampling Method: Non-Probability Sample
Enrollment: 588170 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence and prevalence | 2010 to 2018 fiscal years
  Incidence and prevalence of CKD (by stage), T2DM, and comorbid T2DM/CKD, including 1-, 4-, and 5-year period prevalence and incidence

SECONDARY OUTCOMES:
Comorbidity and complication profiles and rates | 2010 to 2019 fiscal years
  For all three cohorts, comorbidities and complications of interest include:
  1. Diabetic: hypoglycemia, lower limb amputations, diabetic ketoacidosis
  2. Renal: acute kidney injury, acute renal failure, anemia, urogenital tract infections, albuminuria, hematuria, fast estimated glomerular filtration rate decline, CKD progression, continuous renal replacement therapy, dialysis initiation
  3. Cardiovascular: CV events (atrial fibrillation, coronary artery disease, chronic heart failure, hypertension, myocardial infarction, hospitalization for heart failure (specific and broad), peripheral artery disease, stroke/transient ischemic attack (TIA)), CV hospitalization, CV mortality
  4. Other: fractures and all-cause mortality
  5. Any event: Composite outcome to capture any of the above
  For the CKD cohort, results will also be stratified by T2DM status. Comorbidity/complication rates between the T2DM and T2DM/CKD comorbid populations will be compared.
Factors that influence the progression of CKD in patients | 2010 to 2019 fiscal years
  Logistic regression model to assess association of variables of interest (age, sex, health region, comorbidities (Charlson Comorbidity Index as well as conditions in outcome 2), ACR, HbA1c, medication use. This will be performed for all patients with CKD and stratified by T2DM status.
Healthcare resource use (HCRU) and associated costs for CKD patients | 2010 to 2019 fiscal years
  HCRU include: inpatient hospitalizations, hospital length of stay, emergency department visits, general practitioner and specialist visits.
  Costs include: hospital costs, emergency department costs, physician costs, medication costs.
  This will be performed for all patients with CKD and stratified by T2DM status.
Stage-to-stage progression of CKD across the follow-up years in patients with CKD | 2010 to 2019 fiscal years
  This will be performed for all patients with CKD and stratified by T2DM status.
Treatment patterns | 2010 to 2019 fiscal years
  1. Treatment patterns by year for all three cohorts
  2. Drug treatment patterns in patients with T2DM and comorbid CKD versus current guidelines,
  3. Treatment patterns for the CKD cohort will also be stratified by T2DM status.